CLINICAL TRIAL: NCT05196737
Title: Neurophysiological Characterization of Dry Needling in People With Spasticity Due to Stroke--COBRE
Brief Title: DDN in Stroke--COBRE
Acronym: CDN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Gretchen Seif, DPT, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00116575; 5P20GM109040 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-19 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Spasticity, Muscle; CVA
Keywords: Dry Needling; Nervous System; Central Nervous System; Reflexes
MeSH Terms: conditions — Stroke; Muscle Spasticity; Neurologic Manifestations | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All participants completed 2 weeks of the study. Baseline reflex measurements will be collected during the first week of the study (Visits 1-4). No dry needling will occur during this week, with the aim of tracking any natural variability in nervous system excitability at the same time points as reflex measurements during the intervention week. All participants who participated in baseline reflex measurements during week 1 will continue to the second week of the study (Visits 5-7). Participants will receive dry needling to relieve spasticity in the target calf muscle (middle gastrocnemius) during Visit 5. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to DDN, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN. These assessments will examine how you move your leg and how your nervous system responds to non-invasive nerve stimulation.
  Interventions: Behavioral: Dry Needling

INTERVENTIONS:
Behavioral: Dry Needling — Dry needling is a procedure in which a thin, stainless steel needle is inserted into the skin to produce a muscle twitch response. It is intended to release a knot in a muscle and relieve pain.

SUMMARY:
The study team is recruiting 20 adults with spasticity due to chronic stroke for a 7 day study over 2 weeks. In people with chronic stroke, one of the most common and disabling problems is spasticity (increased muscle tone or muscle stiffness). The purpose of this research study is to examine effects of dry needling on the nervous system (pathways between the muscle, spinal cord, and brain) in people with spasticity due to chronic stroke. Dry needling is a procedure in which a thin, stainless steel needle is inserted into the skin to produce a muscle twitch response. It is intended to release a knot in the muscle and relieve pain.

The total study duration is 7 visits over 2 weeks. There will be 4 visits the first week, and 3 visits the second week. The first visit will take about 1.5 hours, during which study staff will determine the best placement of electrodes and create a cast of the participant's leg to aid them in quickly placing the electrodes on the remainder of the visits. The second and fifth visits will last about 3.5 hours, and all other visits will last about 1.5 hours. Dry needling will take place on the fifth visit only. During each visit the participant will be asked to participate in examinations of reflexes (muscle responses to non-invasive nerve stimulation) and leg function.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* no known neurological injuries.
* neurologically stable for >6 months (and >1 yr post stroke)
* medical clearance to participate
* unilateral ankle and/or wrist spasticity, confirmed by Modified Ashworth Scale (MAS) > 1 and the presence of spastic hyperreflexia

Exclusion Criteria:

* motoneuron injury (i.e. the neurons that give rise to the axons innervating the muscles) with inadequate response to stimulation
* a cardiac condition ( history of myocardial infarction, congestive heart failure, pacemaker use, coronary artery disease, atrial fibrillation, congenital heart disease, uncontrolled hypertension)
* a medically unstable condition (including temporary infections and pregnancy)
* age <18 years old
* cognitive impairment sufficient to interfere with informed consent or successful completion of the protocol
* metal allergies
* needle phobias
* lymphedema over a limb (due to risk of infection/cellulitis)
* abnormal bleeding tendencies
* compromised immune system
* vascular disease
* uncontrolled diabetes
* history of epilepsy (as DDN generates strong somatosensory sensation)
* anxiety disorders or in distress
* botox injection in target muscle within 3 months prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Seif, DPT, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in a cross-sectional study. Eleven participants were enrolled in the non-intervention week, of which 9 participants completed all visits. Those 9 participants went on to the Dry Needling Reflex Measurements, of which 8 participants completed all visits. So 11 participants were enrolled, and 8 completed the study procedures.
Groups:
- Non-Intervention Week Reflex Measurements: Baseline reflex measurements will be collected during the first week of the study (Visits 1-4). No dry needling will occur during this week. The aim of this arm is to track any natural variability in nervous system excitability at the same time points as reflex measurements during the intervention week.
Period: Non-intervention Week
Arm/Group | Non-Intervention Week Reflex Measurements
Started | 11
Timepoint 1/Pre-DDN | 9
Timepoint 2/Post Immediate DDN) | 9
Timepoint 3/Post 90 Minutes DDN | 9
Timepoint 4/Post 24 Hours DDN | 9
Timepoint 5/Post 72 Hours DDN | 9
Completed | 9
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Dry Needling Reflex Measurment Week
Arm/Group | Non-Intervention Week Reflex Measurements
Started | 9
Timepoint 1/Pre-DDN | 9
Timepoint 2/Post Immediate DDN) | 9
Timepoint 3/Post 90 Minutes DDN | 9
Timepoint 4/Post 24 Hours DDN | 9
Timepoint 4/Post 24 Hours DDN | 9
Timepoint 5/Post 72 Hours DDN | 8
Completed | 8
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Baseline reflex measurements will be collected during the first week of the study (Visits 1-4). No dry needling will occur during this week. The aim of this arm is to track any natural variability in nervous system excitability at the same time points as reflex measurements during the intervention week.
  All participants who participated in baseline reflex measurements during week 1 will continue to the second week of the study (Visits 5-7). Participants will receive dry needling to relieve spasticity in the target calf muscle (middle gastrocnemius) during Visit 5. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to DDN, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN. These assessments will examine how you move your leg and how your nervous system responds to non-invasive nerve stimulation.
  Dry Needling: Dry needling is a procedure in which a thin, stainless steel needle is inserted into the skin to produce a muscle twitch response. It is intended to release a knot in a muscle and relieve pain.
Arm/Group | Single Arm
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in the H-reflex Amplitude in Response to Nerve Stimulation
Description: H-reflex amplitude (mV) reflects the excitability of its reflex pathway. Changes in the H-reflex amplitude indicate that DDN influences the spinal excitability. This will be measured in the tibialis anterior and the triceps surae.
Time Frame: 7 days prior (2 time points), 6 days prior, 4 days prior, baseline, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN
Population: Due to equipment malfunction, we could not obtain data with adequate quality for this analysis.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Changes in Cutaneous Reflexes Elicited by Non-noxious Stimulation of Cutaneous or Mix Nerves
Description: Changes in the cutaneous reflex amplitudes would indicate that DDN can influence the spinal processing of cutaneous information.
Time Frame: as for outcome 1
Population: Due to equipment malfunction, we could not obtain data with adequate quality for this analysis.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in Perception of Cutaneous Stimuli as Measured by Perception and Radiating Threshold of Cutaneous Nerve Stimulation
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Due to equipment malfunction, we could not obtain data with adequate quality for this analysis.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

4. Primary Outcome: Ability to Move the Limb as Measured by Range of Motion (ROM)
Description: ROM is measured in degrees using a standard goniometer. ROM will be measured both passively (moved by the assessor) and actively (participant moves the leg themselves) and the value reported is the maximum degree of dorsiflexion in each condition. Positive values indicate degrees of dorsiflexion beyond neutral, negative values indicate degrees of plantarflexion. Greater values indicate greater degrees of dorsiflexion.
Time Frame: Timepoints are defined as baseline, 0-minutes post, 90 minutes post and 72 hours post DDN during intervention week and the corresponding 4 timepoints the week prior (non-intervention) but without DDN.
Measure: Median (Standard Deviation); unit: maximum degrees of dorsiflexion
Groups:
- Dry Needling Reflex Measurements: All participants who participated in baseline reflex measurements during week 1 will continue to the second week of the study (Visits 5-7). Participants will receive dry needling to relieve spasticity in the target calf muscle (middle gastrocnemius) during Visit 5. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to DDN, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN. These assessments will examine how you move your leg and how your nervous system responds to non-invasive nerve stimulation.
  Dry Needling: Dry needling is a procedure in which a thin, stainless steel needle is inserted into the skin to produce a muscle twitch response. It is intended to release a knot in a muscle and relieve pain.
Arm/Group | Non-Intervention Week Reflex Measurements | Dry Needling Reflex Measurements
Number analyzed (Participants) | 8 | 8
maximum degrees of dorsiflexion
  passive DF ROM (with knee extended) baseline | 0.5 (4.09) | 0 (3.89)
  passive DF ROM (with knee extended) 0-min post | 0 (4.62) | 0.5 (3.83)
  passive DF ROM (with knee extended) 90-min post | 0 (5.26) | 3 (3.93)
  passive DF ROM (with knee extended) 72 hour post | 0 (6.20) | 0 (11.51)
  active DF ROM (with knee extended) baseline | -28.5 (10.92) | -24.5 (8.94)
  active DF ROM (with knee extended) 0-min post | -26 (11.36) | -22.5 (7.14)
  active DF ROM (with knee extended) 90-min post | -26.5 (9.34) | -22 (9.24)
  active DF ROM (with knee extended) 72-hr post | -22 (11.51) | -21 (12.06)
  passive DF ROM (with knee flexed) baseline | 2.5 (6.00) | 5.5 (5.66)
  passive DF ROM (with knee flexed) post-0 min DDN | 4 (8.30) | 8 (3.70)
  passive DF ROM (with knee flexed) post-90 min DDN | 2.5 (6.57) | 8 (4.93)
  passive DF ROM post-72 hr DDN | 4.5 (4.64) | 5.5 (5.28)
  active DF ROM (with knee flexed) baseline | -24.5 (13.80) | -14 (12.71)
  active DF ROM (with knee flexed) post-0 min DDN | -20 (8.29) | -16 (10.23)
  active DF ROM (with knee flexed) post-90 min DDN | -19 (6.85) | -15.5 (9.52)
  active DF ROM (with knee flexed) post-72 hr DDN | -17 (10.92) | -15.5 (13.15)

5. Secondary Outcome: Ability to Move the Leg as Measured by the Fugl-Meyer Assessment (FMA) Lower Extremity
Description: An increase in the FMA-LE score indicates better movement of the leg. Score ranges from 0 - 34.
Time Frame: as for outcome 4
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Non-Intervention Week\Measurements: Baseline measurements will be collected during the first week of the study (Visits 1-4). No dry needling will occur during this week. The aim of this arm is to track any natural variability in nervous system excitability at the same time points during the intervention week.
- Intervention Week Measurements: All participants who participated in baseline measurements during week 1 will continue to the second week of the study (Visits 5-7). Participants will receive dry needling to relieve spasticity in the target calf muscle (middle gastrocnemius) during Visit 5. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to DDN, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN.
Arm/Group | Non-Intervention Week\Measurements | Intervention Week Measurements
Number analyzed (Participants) | 8 | 8
score on a scale
  Median FMA-LE score baseline | 22 (5.00) | 20 (5.23)
  Median FMA-LE score 0-min post | 24 (5.01) | 19.5 (5.19)
  Median FMA-LE score 90 min post | 22.5 (5.68) | 21 (4.78)
  Median FMA-LE score 72 hr post | 22.5 (5.44) | 21 (4.97)

6. Secondary Outcome: Change in Spasticity as Measured by the Modified Ashworth Scale (mAS)
Description: The mAS score ranges from 0: normal muscle tone to 4: rigid in flexion or extension. A decrease in mAS indicates decreased spasticity. A score of 1.5 reported below is equal to 1+ on the mAS
Time Frame: baseline, immediately after DDN, 90 minutes after DDN, 24 hours after, and 72 hours after DDN
Measure: Number; unit: score on a scale
Groups:
- Baseline: baseline/immediately prior to DDN
- Post-immediate: immediately after DDN
- Post-90 Min: 90 minutes after DDN
- Post-24 Hrs: 24 hours after DDN, single timepoint at this visit
- Post-72 Hrs: 72 hours after DDN, single timepoint at this visit
Arm/Group | Baseline | Post-immediate | Post-90 Min | Post-24 Hrs | Post-72 Hrs
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
score on a scale
  Participant 1 | 3 | 3 | 3 | 3 | 3
  Participant 2 | 3 | 2 | 2 | 2 | 3
  Participant 4 | 2 | 1.5 | 1.5 | 2 | 2
  Participant 5 | 2 | 2 | 2 | 2 | 3
  Participant 6 | 3 | 3 | 3 | 3 | 3
  Participant 8 | 3 | 3 | 3 | 3 | 3
  Participant 14 | 1.5 | 1.5 | 1.5 | 1 | 1

7. Secondary Outcome: Change in Pain Level as Measured by the Visual Analog Scale (VAS) for Pain
Description: Pain is rated by the participant on a scale from 0 (no pain) to 10 (worst pain imaginable). Decreased score on the VAS for pain indicates decreased pain.
Time Frame: as for outcome 1
Population: No pain was reported by any participant throughout the study. All participants reported "0" pain at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 8
score on a scale | 0 (0)

8. Secondary Outcome: Change in Time Needed to Walk 10 Meter (10 m Walk Test)
Description: Decreased time indicates improved ability to walk
Time Frame: Timepoints are defined as baseline, 0-minutes post, 24 hours post and 72 hours post DDN during intervention week and the corresponding 4 timepoints the week prior (non-intervention) but without DDN.
Measure: Median (Standard Deviation); unit: seconds
Groups:
- Non-Intervention Week 10MWT Measurement: Baseline measurements will be collected during the first week of the study (Visits 1-4). No dry needling will occur during this week. The aim of this arm is to track any natural variability in walking speed at the same time points as walking speeds during the intervention week.
- Intervention Week 10MWT Measurement: All participants who participated in baseline measurements during week 1 will continue to the second week of the study (Visits 5-7). Participants will receive dry needling to relieve spasticity in the target calf muscle (middle gastrocnemius) during Visit 5. The study team will examine the effects of this treatment on walking speed by performing assessments just prior to DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN.
Arm/Group | Non-Intervention Week 10MWT Measurement | Intervention Week 10MWT Measurement
Number analyzed (Participants) | 8 | 8
seconds
  Median 10MWT time in seconds at baseline | 9.525 (2.61) | 7.91 (2.25)
  Median 10MWT time in seconds 90 min post | 9.515 (2.52) | 8.1 (2.00)
  Median 10MWT time in seconds 24 hours post | 8.175 (1.99) | 7.57 (2.44)
  Median 10MWT time in seconds 72 hours post | 7.945 (1.90) | 7.555 (2.13)

ADVERSE EVENTS:
Time Frame: 7 days prior, 6 days prior, 4 days prior, baseline, immediately after DDN, 90 minutes after DDN, 24 hours after DDN, and 72 hours after DDN
Description: Each day of participation, study personnel communicated with the participant regarding their general health and any side-effect of the intervention.
Arm/Group | Non-Intervention Week Reflex Measurements | Dry Needling Reflex Measurements
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT05196737/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05196737/ICF_000.pdf